CLINICAL TRIAL: NCT02690584
Title: Metacognitive Therapy for Post-concussive Symptoms After Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1456
Record Dates: First submitted 2016-02-17; First posted 2016-02-24 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Brain Injuries; Post-Concussive Symptom; Post-Concussive Syndrome
Keywords: Psychotherapy
MeSH Terms: conditions — Brain Injuries; Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metacognitive therapy (Experimental): Metacognitive therapy, one 45-60 min session weekly during 10 weeks.
  Interventions: Behavioral: Metacognitive therapy

INTERVENTIONS:
Behavioral: Metacognitive therapy

SUMMARY:
The purpose of this open trial is to investigate the feasibility, acceptability, and effect of metacognitive therapy in patients with prolonged post-concussive symptoms after mild traumatic brain injury.

ELIGIBILITY:
Patients with prolonged recovery after mild TBI (GCS >12) will be recruited to our study if they have post concussive symptoms > 6 months after injury.

Patients will be recruited from an ongoing cohort study investigating mild and moderate TBI at St. Olavs Hospital and Trondheim Municipality Emergency Clinic, and in addition (as of October 2017) among TBI patients at St Olavs Hospital who were not included in the cohort study.

Inclusion criteria

* Aged ≥between 16 and < 60 years
* Have sustained a traumatic brain injury

Exclusion criteria

* Severe TBI (GCS score 8 or less)
* Non fluency in Norwegian
* Living outside of Norway
* Major other trauma with high risk of disability lasting more than 3 months.
* Major incidental intracranial findings in acute MRI e.g. cyst, tumor, malformation, infarctions.
* Severe psychiatric, neurological or medical disease, including: Psychotic disorders, bipolar disorder, ongoing severe depressive episode

  * Personality disorders affecting adherence to the research protocol
  * Alcohol/drug abuse affecting adherence to the research protocol
  * Mental retardation, autism or other severe developmental disorders
  * Prior complicated mild, moderate or severe TBI
  * Stroke or other acquired brain injuries
  * Progressive neurological disorders (e.g. Parkinson's disease, MS)
  * Advanced cancer, heart- or respiratory disease or other somatic diseases that interfere with function.
  * Major other trauma e.g. spinal cord injury

In addition to exclusion criteria already employed in the cohort study, patients with co-occurring psychiatric disorders that necessitate referral to specific treatment according to existing guidelines will be excluded from the current intervention study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
symptoms assessed by Rivermead Post Concussion Symptoms Questionnaire | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after completed therapy

SECONDARY OUTCOMES:
Conners CPT-III | 2 pre-treatment baseline measures, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
D-KEFS Trail Making Test | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Color-Word Interference Test | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
D-KEFS Verbal Fluency | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Symbol Digit Modality Test | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Behavior Rating Inventory-Adult version (BRIEF-A) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
The metacognitive beliefs questionnaire (MCQ-30) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Fatigue questionnaire (FQ) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Brief Pain Inventory (BPI) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Inventory of Interpersonal Problems 64 (IIP-64) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Fatigue severity scale (FSS) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
SF-12 | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Resilience scale for Adults (RSA) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Epworth sleepiness scale (ESS) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Insomnia severity Index (ISI) | baseline, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Beck Depression Inventory (BDI) | 3 pre-treatment baseline measures, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Beck Anxiety Inventory (BAI) | 3 pre-treatment baseline measures, immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy
Cognitive Attention Syndrome (CAS-1) | 3 pre-treatment baseline measures, session to session (10 sessions), immediately after last therapy session, 10 weeks after completed therapy, 6 months after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Magne Arve Flaten, phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Psykologisk Institutt, Dragvoll, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided